CLINICAL TRIAL: NCT02395185
Title: A Randomized Controlled Trial of Three Non-pharmacologic Analgesic Techniques for Casting of Clubfoot Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: Kosair Charities, Inc. (Other); University of Kentucky (Other)
Responsible Party: Principal Investigator, Todd Milbrandt, MD, Shriners Hospitals for Children
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: LEX-102
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-05

CONDITIONS: Clubfoot
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Milk (Experimental): Milk bottle administration
  Interventions: Other: Milk bottle administration; Other: Water bottle administration; Other: Sucrose bottle administration
- Water (Experimental): Water bottle administration
  Interventions: Other: Milk bottle administration; Other: Water bottle administration; Other: Sucrose bottle administration
- Sucrose (Experimental): Sucrose bottle administration
  Interventions: Other: Milk bottle administration; Other: Water bottle administration; Other: Sucrose bottle administration

INTERVENTIONS:
Other: Milk bottle administration — Patients are given a bottle of milk during the casting process.
Other: Water bottle administration — Patients are given a bottle of water during the casting process.
Other: Sucrose bottle administration — Patients are given a bottle of sucrose during the casting process.

SUMMARY:
While it has been shown that sucrose or milk ingestion decreases pain responses in heel sticks, no study up to this point has determined the best intervention for decreasing the pain response during casting for clubfoot deformity.

The goal of this study is to investigate the effect of three different non-pharmacologic interventions (sucrose, milk, water) on pain response during clubfoot casting.

This study will allow us to discern the best non-pharmacologic intervention for pain control during clubfoot casting and to provide a more pleasant, comfortable experience for patients and families.

DETAILED DESCRIPTION:
Clubfoot deformity in newborns is common, occurring in 1-2/1000 births. Treatment of this deformity has shifted from surgical to non-surgical management. The non-surgical management includes utilizing the Ponseti technique of manipulation and casting, followed by Achilles tenotomy and brace application. The newborn undergoes, on average, 4-6 casts before the foot deformity is corrected. During this manipulation and casting, the infants can become fussy and irritable. This irritability is likely due to discomfort felt from the manipulative process and subsequent casting.

Studies that have focused on decreasing the pain response to heel sticks for laboratory testing in the neonatal intensive care units used sucrose or milk ingestion and swaddling in newborns to decrease pain responses. Both sucrose and milk have been shown to decrease the pain response as measured by the Premature Infant Pain Profile (PIPP) or the Bernese Pain Scale for Neonates. In addition, other pain scales have been used in newborn babies including the CRIES, CHIPPS, NIPS, and COMFORT scales to evaluate the effectiveness of pain relieving interventions. These scales were used alongside objective physiologic measurements such as heart rate, heart rate variability (HRV), respiratory rate, and oxygen saturation.

While it has been shown that sucrose or milk ingestion decreases pain responses in heel sticks, no study up to this point has determined the best intervention for decreasing the pain response during casting for clubfoot deformity. The goal of this study is to investigate the effect of three different non-pharmacologic interventions (sucrose, milk, water) on pain response during clubfoot casting, allowing us to discern the best non-pharmacologic intervention for pain control during clubfoot casting and to provide a more pleasant, comfortable experience for patients and families. A secondary objective is to investigate whether or not family environment or the level of anxiety felt by the parents impacts the pain felt by the infant during the casting process.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic clubfoot deformity
* undergoing clubfoot casting for correction

Exclusion Criteria:

* cannot use a bottle for feeding
* on solid food
* have had surgery
* have been given an analgesic within three hours prior to data collection

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd M Milbrandt, MD, Principal Investigator — Shriners Hospital for Children, Mayo Clinic

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 53 participants were assessed for eligability. 33 patient participants and their guardians were enrolled in the study from 3/13/13 to 9/17/14 at their initial clinical visit. A total of 131 casts were performed.
Groups:
- All Participants: 33 Participants were randomized to one of 18 sequences of milk, water, or formula for an average of 6 casting visits.
Period: Overall Study
Arm/Group | All Participants
Started | 33 (32 guardians participated with these infants. one infant did not have a guardian participate.)
Sequence 1 (s,s,m,m,w,w) | 2 (one of the participants in this milestone did not have a guardian enrolled due to age.)
Sequence 2 (w,s,s,m,m,w) | 2
Sequence 3 (w,w,s,s,m,m) | 2
Sequence 4 (m,w,w,s,s,m) | 2
Sequence 5 (m,m,w,w,s,s) | 2
Sequence 6 (s,m,m,w,w,s) | 2
Sequence 7 (s,s,w,w,m,m) | 2
Sequence 8 (m,s,s,w,w,m) | 2
Sequence 9 (m,m,s,s,w,w) | 2
Sequence 10 (w,m,m,s,s,w) | 2
Sequence 11 (w,w,m,m,s,s) | 2
Sequence 12 (s,w,w,m,m,s) | 2
Sequence 13 (s,m,w,m,s,w) | 2
Sequence 14 (w,s,m,w,m,s) | 2
Sequence 15 (s,w,s,m,w,m) | 2
Sequence 16 (m,s,w,s,m,w) | 1
Sequence 17 (w,m,s,w,s,m) | 1
Sequence 18 (m,w,m,s,w,s) | 1
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis included 43 casts receiving sucrose, 37 casts receiving milk or formula, and 42 casts receiving water
Groups:
- All Participants: Bottle Administration: 2 oz of sucrose, water, or milk/formula given in a bottle during the casting process
  Bottle Administration: Patients are given a bottle during the casting process. Contents of bottle depend on the arm to which they are randomized.
Arm/Group | All Participants
Number analyzed (Participants) | 33
Age, Customized [Number; unit: participants]
  <=18 years | 33
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 17.9 (20.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: NIPS (Neonatal Infant Pain Scale)
Description: Each cast visit will be videotaped before, during, and after casting, and later reviewed for subjective evaluation of pain using NIPS (Neonatal Infant Pain Scale). The NIPS examines six behavioral groupings that contribute to a pain score ranging from 0 to 7: facial expression (relaxed muscles or grimace), cry (no cry, whimper, or vigorous cry), breathing patterns (relaxed, change in breathing), arms (relaxed/restrained, flexed/extended), legs (relaxed/restrained, flexed/extended), state of arousal (sleeping/awake, fussy). Scoring will take place by a trained study personnel blinded to the contents of the bottle. Scoring for all measures will be recorded at minute intervals. A pre casting score from the average of the first 3 minute scores prior to casting; a during casting score from the average of the scores at 1 minute intervals during casting; and a post casting score from the average of the 3 minute scores post casting. Scores are categorized as 0 no pain, to >4 severe pain.
Time Frame: Scoring will be recorded at minute intervals starting at 2 minutes prior to casting and ending at 3 minutes post casting.
Population: Because this was a crossover design, multiple casts were assessed for each participant
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: casts
Groups:
- Milk: Bottle Administration: 2 oz milk or formula given in a bottle during the casting process
  Bottle Administration: Patients are given a bottle during the casting process. Contents of bottle depend on the arm to which they are randomized.
- Water: Bottle Administration: 2 oz water given in a bottle during the casting process
  Bottle Administration: Patients are given a bottle during the casting process. Contents of bottle depend on the arm to which they are randomized.
- Sucrose: Bottle Administration: 2 oz sucrose solution given in a bottle during the casting process
  Bottle Administration: Patients are given a bottle during the casting process. Contents of bottle depend on the arm to which they are randomized.
Arm/Group | Milk | Water | Sucrose
Number analyzed (Participants) | 24 | 26 | 29
Number analyzed (casts) | 37 | 39 | 43
units on a scale
  NIPS pre casting | 2.28 (2.38) | 1.63 (2.12) | 1.84 (2.18)
  NIPS casting | 0.91 (1.26) | 2.22 (2.01) | 0.63 (1.27)
  NIPS post casting | 2.11 (2.37) | 1.49 (2.29) | 0.69 (1.53)

2. Secondary Outcome: Heart Rate
Description: Heart rate will be recorded at minute intervals. A pre casting measure from the average of the first 3 minute measures prior to casting; a during casting measure from the average of the measures at 1 minute intervals during casting; and a post casting measure from the average of the 3 minute measures post casting.
Time Frame: Heart rate will be recorded at minute intervals starting at 2 minutes prior to casting and ending at 3 minutes post casting.
Population: Because this was a crossover design, multiple casts were assessed for each participant
Measure: Mean (Standard Deviation); unit: bpm
Units Other Than Participants: casts
Arm/Group | Milk | Water | Sucrose
Number analyzed (Participants) | 24 | 26 | 29
Number analyzed (casts) | 37 | 39 | 43
bpm
  pre casting | 152.72 (20.45) | 145.69 (17.12) | 155.9 (15.71)
  casting | 152.54 (12.87) | 152.59 (9.03) | 154.33 (24.55)
  post casting | 147.2 (12.05) | 143.89 (13.06) | 149.78 (12.99)

3. Secondary Outcome: Oxygen Saturation
Description: Oxygen saturation will be recorded at minute intervals. A pre casting measure from the average of the first 3 minute measures prior to casting; a during casting measure from the average of the measures at 1 minute intervals during casting; and a post casting measure from the average of the 3 minute measures post casting.
Time Frame: Oxygen saturation will be recorded at minute intervals starting at 2 minutes prior to casting and ending at 3 minutes post casting
Population: Because this was a crossover design, multiple casts were assessed for each participant
Measure: Mean (Standard Deviation); unit: percentage of SpO2
Units Other Than Participants: casts
Arm/Group | Milk | Water | Sucrose
Number analyzed (Participants) | 24 | 26 | 29
Number analyzed (casts) | 37 | 39 | 43
percentage of SpO2
  pre casting | 98 (1.57) | 97.52 (2.26) | 98.33 (1.63)
  casting | 97.38 (1.26) | 97.56 (3.23) | 94.32 (12.43)
  post casting | 98.07 (2.07) | 97.85 (2.34) | 98.18 (1.62)

ADVERSE EVENTS:
Time Frame: up to four weeks after study participation
Description: Patients were monitored for gastrointestinal, systemic, or allergic reactions during routine clinical follow-up visits.
Groups:
- Milk or Formula: Bottle Administration: 2 oz milk or formula given in a bottle during the casting process
  Bottle Administration: Patients are given a bottle during the casting process. Contents of bottle depend on the arm to which they are randomized.
Arm/Group | Sucrose | Milk or Formula | Water
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 1/29 | 0/26 | 0/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sucrose (N=29) | Milk or Formula (N=26) | Water (N=26)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — At 7 days post-treatment, subject's guardian reported that the subject was gassy, spitt up, didn't eat well, and diarrhea with chapped bottom following treatment but that the problem had resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No